CLINICAL TRIAL: NCT05741684
Title: Combining Internet-Delivered Cognitive Behavioral Therapy and Attention Bias Modification for Depression in Firefighters
Brief Title: iCBT and ABM for Reducing Depressive Symptoms in Firefighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adai Technology (Beijing) Co., Ltd. (Other)
Collaborators: Kungming Training Corps of National Fire and Rescue Administration (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XF001
Record Dates: First submitted 2023-02-12; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCBT and ABM (Experimental): A combined internet-delivered Cognitive Behavioral Therapy (iCBT) and Attention Bias Modification (ABM) intervention to reduce depressive symptoms in firefighters.
  Interventions: Behavioral: Internet-delivered Cognitive Behavioral Therapy; Behavioral: Attention Bias Modification
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Internet-delivered Cognitive Behavioral Therapy — iCBT was administered in an unguided fashion without human therapeutic support. Participants were instructed to progress through the eight core modules over an 8-week period. The modules comprised psychoeducational content centered around CBT, aimed at promoting the development of skills such as self-monitoring of emotions, cognitive distancing, cognitive reframing/restructuring, problem-solving, and mindfulness. In the event of technical difficulties during the intervention, participants were able to seek assistance.
  Arms: iCBT and ABM
Behavioral: Attention Bias Modification — The Dot-Probe Paradigm was utilized within the Attention Bias Modification procedure. The training sessions were comprised of 96 trials, which included facial expression photos depicting happiness, neutrality, and sadness, sourced from four male and four female actors. A fixed cross (+) was presented on the computer screen's center for a duration of 500 milliseconds before each stimulus display, followed by the presentation of two images portraying distinct emotional expressions, which persisted for 500 milliseconds. After the disappearance of the images, an arrow appeared in the location where they had been displayed, and participants were instructed to select the arrow that corresponded with the presented arrow. In the ABM procedure, the arrow was consistently presented following the display of a more positive facial expression, such that in the instance of a sad-neutral face pair, the arrow would always appear in the location of the neutral facial expression image.
  Arms: iCBT and ABM

SUMMARY:
The study aimed to examine the impact of a combined internet-delivered Cognitive Behavioral Therapy (iCBT) and Attention Bias Modification (ABM) intervention to reduce depressive symptoms in firefighters. The study was a randomized controlled trial carried out in Kunming, China, and involved the recruitment of 138 active firefighters as participants. The intervention lasted for an 8-week duration, during which participants participated in ABM exercises on alternating days and concurrently underwent four modules of iCBT courses delivered through a smartphone application.

ELIGIBILITY:
Inclusion Criteria:

* being an active firefighter and aged between 18 and 50
* having a score greater than zero on the Patient Health Questionnaire-9 (PHQ-9)
* with no history of severe depression

Exclusion Criteria:

* having suicidal ideation or intent
* having an active psychotic disorder other than depression
* prior participation in a cognitive-behavioral intervention
* concurrent participation in another study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 | Baseline
  The Patient Health Questionnaire-9 (PHQ-9) was utilized to assess symptoms of depression. The PHQ-9 is a self-report questionnaire comprising 9 items, with a score range of 0-27, measuring depression-related symptoms experienced in the past two weeks
Patient Health Questionnaire-9 | Immediately Post-intervention
  The Patient Health Questionnaire-9 (PHQ-9) was utilized to assess symptoms of depression. The PHQ-9 is a self-report questionnaire comprising 9 items, with a score range of 0-27, measuring depression-related symptoms experienced in the past two weeks
Attention Bias Score | Baseline
  To quantify attention bias, response times (RTs) were analyzed in accordance with the established procedure to calculate the attention bias score (ABS). Trials characterized by inaccurate responses or RTs of exceptional brevity (<150ms) or prolonged duration (>1200ms) were disregarded. The computation of attention bias entailed determining the discrepancy between the mean RT in response to relatively positive stimuli and the mean RT in response to relatively negative stimuli. A preference for happy faces was indicated by an average RT for happy facial expressions that were shorter than the average RT for neutral or sad facial expressions.
Attention Bias Score | Immediately Post-intervention
  To quantify attention bias, response times (RTs) were analyzed in accordance with the established procedure to calculate the attention bias score (ABS). Trials characterized by inaccurate responses or RTs of exceptional brevity (<150ms) or prolonged duration (>1200ms) were disregarded. The computation of attention bias entailed determining the discrepancy between the mean RT in response to relatively positive stimuli and the mean RT in response to relatively negative stimuli. A preference for happy faces was indicated by an average RT for happy facial expressions that were shorter than the average RT for neutral or sad facial expressions.
Attention Bias Variability | Baseline
  To quantify attention-bias variability (ABV), the experimental data were divided into 8 segments, and attention-bias scores were computed for each segment. Subsequently, the standard deviation of attention-bias scores across segments was determined, and this value was divided by all trials ABS to account for ABS variability.
Attention Bias Variability | Immediately Post-intervention
  To quantify attention-bias variability (ABV), the experimental data were divided into 8 segments, and attention-bias scores were computed for each segment. Subsequently, the standard deviation of attention-bias scores across segments was determined, and this value was divided by all trials ABS to account for ABS variability.

CONTACTS AND LOCATIONS:
Locations (1):
- Kunming Training Corps of the National Fire and Rescue Administration, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No
Data not available due to privacy and ethical considerations